CLINICAL TRIAL: NCT03140787
Title: Assessment of Efficacy and Safety of Primary Maxillary Second Molars Anesthesia Using Nasal Spray in Children
Brief Title: Efficacy and Safety of Primary Teeth Anesthesia Using Nasal Spray in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Pedo-01-2017
Record Dates: First submitted 2017-04-14; First posted 2017-05-04 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Spray of Lidocaine HCL (Experimental): This group will receive treatment with an application of nasal spray for anesthetization.
  Interventions: Drug: Nasal Spray of Lidocaine HCL
- Infiltration injection of Lidocaine HCL (Active Comparator): Each patient in this group will receive an infiltration injection for anesthetization
  Interventions: Drug: Infiltration injection of Lidocaine HCL

INTERVENTIONS:
Drug: Nasal Spray of Lidocaine HCL — This spray consists of lidocaine hydrochloride-epinephrine hydrochloride
  Arms: Nasal Spray of Lidocaine HCL
Drug: Infiltration injection of Lidocaine HCL — This is the ordinary method of establishing anesthesia for patients undergoing dental treatment for caries.
  Arms: Infiltration injection of Lidocaine HCL

SUMMARY:
68 healthy children from the Department of Pediatric Dentistry at Damascus University who require treatment for their primary maxillary second molars will be randomly assigned into one of two groups: experimental or control groups. In the experimental group, a lidocaine hydrochloride-epinephrine hydrochloride nasal spray will be applied to anesthetize upper second molar before the commencement of treatment.

To assess the efficacy of this kind of anesthesia, a specific scale will be used by an external observer after capturing some video files of the performed treatment.

To assess the safety of this procedure, vital signs will be recorded before and after treatment.

Acceptance of the nasal spray will be recorded based on the child's behavior before and after treatment using Frankl scale.

If anesthesia was not sufficient to proceed with the procedure, a rescue anesthesia would be used. Rescue anesthesia consists of an infiltration injection of lidocain hydrochloride 2% with epinephrine hydrochloride (1:100,000). In the control group, an intra-oral lidocaine-epinephrine injection will be applied due to treatment. Safety, efficacy and acceptance will be assessed in the same manner to what is performed in the experimental group.

DETAILED DESCRIPTION:
The most common method for anesthetizing maxillary teeth is infiltration injection of an anesthetic agent. This approach carries several disadvantages. First is the child's fear of pain. Infection is also a risk for providers, through exposure to blood-borne pathogens via needle stick.

Fear of a painful dental injection and subsequent avoidance behavior are significant barriers to regular visits to the dentist.

Importantly, patients' fear of injections can delay needed dental care. Surveys indicate that 30-40 million people in the US avoid going to the dentist because of fear of pain and anesthetic injections.

Therefore an anesthetic procedure that would avoid the discomfort of a local anesthetic injection thus obviating fear and anxiety about receiving a "shot," would greatly benefit dental patients. Further, for procedures involving more than one maxillary tooth on the same side, a trans-nasally applied anesthetic agent that could anesthetize multiple maxillary teeth at once instead of use of repeated infiltration injections would be a major convenience for patients and dentists.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children between 7-10 years.
2. With a need for pulpotomy or a restorative dental procedure requiring local anesthesia for a single vital primary maxillary second molar with no evidence of pulpal necrosis.
3. Normal lip, nose, eyelid, and cheek sensation.
4. No history of allergy for lidocaine-hydrochloride or epinephrine-hydrochloride.

Exclusion Criteria:

1. Frequent bleeding form the nose (≥ 5 per month)
2. Inadequately controlled active thyroid disease of any type.
3. Having received dental care requiring a local anesthetic within the 24 hours preceding study entry.
4. History of allergy to or intolerance of lidocaine or epinephrine.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure | (1) five minutes before drug administration, (2) after 10 minutes of anesthesia, and (3) at the completion of the dental treatment, an average of 40 minutes.
  Systolic and diastolic blood pressure will be measured.
Change in Oxygen Saturation | (1) five minutes before drug administration, (2) after 10 minutes of anesthesia, and (3) at the completion of the dental treatment, an average of 40 minutes.
  Oxygen saturation will be measured using a specific device.
Change in Respiration Rate | (1) five minutes before drug administration, (2) after 10 minutes of anesthesia, and (3) at the completion of the dental treatment, an average of 40 minutes.
  Respiration rate will be measured clinically in the conventional manner.
Change in Heart Pulse Rate | (1) five minutes before drug administration, (2) after 10 minutes of anesthesia, and (3) at the completion of the dental treatment, an average of 40 minutes.
  Heart pulse rate will be measured clinically in the conventional manner.
Change in FLACC scale | (1) within the first minute of drug administration, (2) when probing the gingiva at approx. Minute 5, (3) when entering the dentin at approx. Minute 10, (4) when exposing the pulp at approx. Minute 15, (5) during the removal of the pulp at Minute 20
  This scale will be used to evaluate efficacy. It will be studied by an external observer at 5 stages; first stage: during administration of the drug, second stage: while probing the gingiva around the tooth "buccally, palatally", third stage: when penetration of the dentino-enamel junction occurs, fourth stage: when exposure of the dental pulp occurs, fifth stage: during the removal of the coronal pulp.
Change in Frankl scale | (1) within the first minute of drug administration, (2) when probing the gingiva at approx. Minute 5, (3) when entering the dentin at approx. Minute 10, (4) when exposing the pulp at approx. Minute 15, (5) during the removal of the pulp at Minute 20
  This scale will be used to evaluate children's acceptance and will be measured by an external observer at five assessment times.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Raslan Alzein, DDS, Principal Investigator — MSc student, Department of Paedodontics, University of Damascus Dental School; Shadi Azzawi, DDS MSc PhD, Study Director — Senior Lecturer in Paedodontics, Department of Paedodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Peadodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciancio SG, Hutcheson MC, Ayoub F, Pantera EA Jr, Pantera CT, Garlapo DA, Sobieraj BD, Almubarak SA. Safety and efficacy of a novel nasal spray for maxillary dental anesthesia. J Dent Res. 2013 Jul;92(7 Suppl):43S-8S. doi: 10.1177/0022034513484334. Epub 2013 May 20. PMID 23690356
- [Background] Reed KL, Malamed SF, Fonner AM. Local anesthesia part 2: technical considerations. Anesth Prog. 2012 Fall;59(3):127-36; quiz 137. doi: 10.2344/0003-3006-59.3.127. PMID 23050753
- [Background] Pandey RK, Bahetwar SK, Saksena AK, Chandra G. A comparative evaluation of drops versus atomized administration of intranasal ketamine for the procedural sedation of young uncooperative pediatric dental patients: a prospective crossover trial. J Clin Pediatr Dent. 2011 Fall;36(1):79-84. doi: 10.17796/jcpd.36.1.1774746504g28656. PMID 22900449
- [Background] Hersh EV, Pinto A, Saraghi M, Saleh N, Pulaski L, Gordon SM, Barnes D, Kaplowitz G, Bloom I, Sabti M, Moore PA, Lee S, Meharry M, He DY, Li Y. Double-masked, randomized, placebo-controlled study to evaluate the efficacy and tolerability of intranasal K305 (3% tetracaine plus 0.05% oxymetazoline) in anesthetizing maxillary teeth. J Am Dent Assoc. 2016 Apr;147(4):278-87. doi: 10.1016/j.adaj.2015.12.008. Epub 2016 Jan 25. PMID 26822100
- [Background] Kanaa MD, Whitworth JM, Meechan JG. A comparison of the efficacy of 4% articaine with 1:100,000 epinephrine and 2% lidocaine with 1:80,000 epinephrine in achieving pulpal anesthesia in maxillary teeth with irreversible pulpitis. J Endod. 2012 Mar;38(3):279-82. doi: 10.1016/j.joen.2011.11.010. Epub 2011 Dec 22. PMID 22341059
- [Background] Kanaa MD, Whitworth JM, Meechan JG. A prospective randomized trial of different supplementary local anesthetic techniques after failure of inferior alveolar nerve block in patients with irreversible pulpitis in mandibular teeth. J Endod. 2012 Apr;38(4):421-5. doi: 10.1016/j.joen.2011.12.006. Epub 2012 Feb 2. PMID 22414822